CLINICAL TRIAL: NCT01632241
Title: A Phase 3/4, Multi-Center, Randomized, Double-Blind, Placebo-Controlled, 52-Week Study to Evaluate the Efficacy and Safety of Belimumab (HGS1006) in Adult Subjects of Black Race With Systemic Lupus Erythematosus (SLE)
Brief Title: Efficacy and Safety of Belimumab in Black Race Patients With Systemic Lupus Erythematosus (SLE)
Acronym: EMBRACE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Human Genome Sciences Inc., a GSK Company (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Organization: GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 115471; HGS1006-C1112 (Other: Human Genome Sciences Inc.); 2011-005672-42 (EudraCT Number); U1111-1139-9723 (Other: Universal Trial Number)
Record Dates: First submitted 2012-06-28; First posted 2012-07-02 (Estimated); Results first posted 2019-07-05 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-08

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Systemic Lupus Erythematosus; African Continental Ancestry Group; Autoimmune Disease; Antibodies; Minority Groups; Black Race; African Americans; SLE; Belimumab; Lupus
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Autoimmune Diseases | interventions — Standard of Care; belimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo plus standard therapy (Placebo Comparator): Placebo IV plus standard therapy; placebo administered on Days 0, 14, 28, and every 28 days thereafter through Week 48, with a final evaluation at Week 52 in the double-blind period. In the open-label extension period, placebo patients who opt to participate will receive belimumab 10 mg/kilogram (kg) IV every 28 days for an additional 6 months.
  Interventions: Biological: Placebo plus standard therapy; Drug: Standard therapy
- Belimumab 10 mg/kg plus standard therapy (Experimental): Belimumab 10 mg/kg IV plus standard therapy; belimumab administered on Days 0, 14, 28, and then every 28 days thereafter through Week 48, with a final evaluation at Week 52 in the double-blind period. In the open-label extension period, patients who opt to participate will continue to receive belimumab 10 mg/kg IV every 28 days for an additional 6 months.
  Interventions: Biological: Belimumab 10 mg/kg plus standard therapy; Drug: Standard therapy

INTERVENTIONS:
Biological: Placebo plus standard therapy — Placebo plus standard therapy
  Arms: Placebo plus standard therapy
Biological: Belimumab 10 mg/kg plus standard therapy — Belimumab 10mg/kg plus standard therapy
  Arms: Belimumab 10 mg/kg plus standard therapy
Drug: Standard therapy — Standard therapy comprises any of the following (alone or in combination): corticosteroids, antimalarials, non-steroidal anti-inflammatory drugs (NSAIDs), and immunosuppressives; biologics and intravenous cyclophosphamide are not permitted.

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety, and tolerability of belimumab in adult patients of black race with systemic lupus erythematosus (SLE; lupus).

DETAILED DESCRIPTION:
Study participants receive stable standard therapy for lupus in addition to receiving either placebo (no active medicine) or belimumab. The controlled period of the study is 52 weeks. The random assignment in this study is "2 to 1" which means that for every 3 participants, 2 will receive belimumab and 1 will receive placebo. Participants who successfully complete the 52-week study may enter into a 6-month open-label extension. All participants in the open-label extension receive belimumab plus standard therapy.

ELIGIBILITY:
Inclusion criteria:

* At least 18 years of age.
* Self-identified black race.
* Have a clinical diagnosis of SLE according to the American College of Rheumatology (ACR) criteria
* Have active SLE disease defined as a SELENA SLEDAI score >= 8 at screening
* Have 2 unequivocally positive autoantibody test results defined as a positive antinuclear antibody (ANA) test [i.e., titer >= 1:80 by human epithelial cell line 2 (HEp-2) immunofluorescence assay (IFA) and/or positive enzyme immunoassay (EIA)] and/or a positive anti- double stranded deoxyribonucleic acid (dsDNA) (>= 30 international units [IU]/milliliter [mL]) serum antibody test as follows:

  * From 2 independent time points within the study screening period. Screening results must be based on the study's central laboratory results, OR
  * One positive historical test result and 1 positive test result during the screening period.

Historical documentation of a positive ANA test (e.g., HEp-2 IFA or EIA) or anti-dsDNA (eg, anti-dsDNA by any validated commercial assay) must include the date and type of the test, the name of the testing laboratory, numerical reference range, and a key that explains values provided as positive versus negative OR negative, equivocal/borderline positive). Only unequivocally positive values as defined in the laboratory's reference range are acceptable; borderline values will not be accepted.

* On a stable SLE treatment regimen consisting of any of the following medications (alone or in combination) for a period of at least 30 days prior to Day 0 (i.e., day of 1st dose of study agent):

  * Corticosteroids (prednisone or prednisone equivalent, up to 40 mg/day): For subjects on SLE combination therapy, their stable steroid dose must be fixed within the range of 0 to 40 mg/day (prednisone or prednisone equivalent). For subjects whose only SLE treatment is steroids, their stable steroid dose must be fixed within the range of 7.5 to 40 mg/day (prednisone or prednisone equivalent). For those subjects on alternating day doses of steroids, use the average of 2 daily doses to calculate the average daily steroid dose.
  * Other immunosuppressive or immunomodulatory agents including methotrexate, azathioprine, leflunomide, mycophenolate (including mycophenolate mofetil, mycophenolate mofetil hydrochloride, and mycophenolate sodium), calcineurin inhibitors (e.g., tacrolimus, cyclosporine), sirolimus, oral cyclophosphamide, 6-mercaptopurine, mizoribine, or thalidomide.
  * Anti-malarials (e.g., hydroxychloroquine, chloroquine, quinacrine).
  * Non-steroidal anti-inflammatory drugs (NSAIDs).

Note:

* Pre-existing SLE medications must be stable for at least 30 days prior to Day 0.
* Corticosteroids may be added as new medication or their doses adjusted only up to 30 days prior to Day 0.
* New SLE therapy other than corticosteroids must not be added within 60 days of Day 0.
* A female subject is eligible to enter the study if she is:

  * Not pregnant or nursing;
  * Of non-childbearing potential defined as: pre-menopausal females with a documented tubal ligation, hysterectomy, documented hysteroscopic tubal occlusion procedure with follow-up confirmation of bilateral tubal occlusion, or documented bilateral oophorectomy, OR postmenopausal defined as 12 months of spontaneous amenorrhea with an appropriate clinical profile [e.g., > 45 years, in the absence of hormone replacement therapy or other cause for amenorrhea]; in questionable cases obtain a blood sample for follicle stimulating hormone (FSH) and estradiol simultaneously to confirm. Diagnostic levels for FSH and estradiol vary by specific laboratories/assays;
  * OR is of child-bearing potential with negative pregnancy test as determined by serum human chorionic gonadotrophin (hCG) test at screening and urine hCG test prior to dosing AND agrees to use one of the contraception methods for 2 weeks prior to the day of dosing to sufficiently minimize the risk of pregnancy at that point. Female subjects must agree to use contraception until 16 weeks following the last dose of study agent.
  * OR has only same-sex partners, when this is her preferred and usual lifestyle.
  * Have the ability to understand the requirements of the study, provide written informed consent (including consent for the use and disclosure of research-related health information), and comply with the study protocol procedures (including required study visits).

Exclusion criteria:

* Have received treatment with anti-B lymphocyte stimulator (BLyS) [belimumab] at any time.
* Have received any of the following within 364 days of Day 0:

  * Abatacept
  * Other B cell targeted therapy (e.g., rituximab, other anti-cluster of differentiation [CD] 20 agents, anti-CD22 [epratuzumab], anti-CD52 [alemtuzumab], BLyS-receptor fusion protein [BR3], TACI-Fc, or anti-B-cell activating factor [BAFF] (LY2127399).
  * A biologic investigational agent other than B cell targeted therapy (e.g., abetimus sodium, anti-CD40L antibody [BG9588/IDEC-131]).
* Have required 3 or more courses of systemic corticosteroids for concomitant conditions (e.g., asthma, atopic dermatitis) within 364 days of Day 0. (Topical or inhaled steroids are permitted.)
* Have received any of the following within 90 days of Day 0:

  * Anti-tumor necrosis factor (TNF) therapy (eg, adalimumab, certolizumab pegol, etanercept, golimumab, infliximab).
  * Intravenous (IV) cyclophosphamide
  * Interleukin-1 receptor antagonist (anakinra).
  * Intravenous immunoglobulin (IVIG).
  * High dose prednisone or equivalent (> 100 mg/day).
  * Plasmapheresis.
* Have received any of the following within 60 days of Day 0:

  * A non-biologic investigational agent.
  * Any new immunosuppressive/immunomodulatory agent, anti-malarial, or NSAID Note: New inhaled and topical steroids and new topical immunosuppressive agents (e.g., eye drops, topical creams) are allowed. Any NSAID use for < 1 week is allowed.
  * Any steroid injection (e.g., intramuscular, intraarticular, or intravenous).
* Have received any of the following within 30 days of Day 0:

  * A live vaccine.
  * A change in dose of a corticosteroid, other immunosuppressive/immunomodulatory agent, anti-malarial, or NSAID
* Have severe lupus kidney disease (defined by proteinuria > 6 grams/24 hour or equivalent using spot urine protein to creatinine ratio, or serum creatinine > 2.5 mg/deciliter [dL]), or have severe active nephritis requiring acute therapy not permitted by protocol (e.g., IV cyclophosphamide within 90 days of Day 0), or have required hemodialysis or high-dose prednisone (> 100 mg/day) within 90 days of Day 0.
* Have severe active central nervous system (CNS) lupus (including seizures, psychosis, organic brain syndrome, cerebrovascular accident [CVA], cerebritis, or CNS vasculitis) requiring therapeutic intervention within 60 days of Day 0.
* Have a history of a major organ transplant (e.g., heart, lung, kidney, liver) or hematopoietic stem cell/marrow transplant.
* Have clinical evidence of significant unstable or uncontrolled acute or chronic diseases not due to SLE (i.e., cardiovascular, pulmonary, hematologic, gastrointestinal, hepatic, renal, neurological, malignancy, or infectious diseases) which, in the opinion of the principal investigator, could confound the results of the study or put the subject at undue risk.
* Have a planned surgical procedure or a history of any other medical disease (e.g., cardiopulmonary), laboratory abnormality, or condition (e.g., poor venous access) that, in the opinion of the principal investigator, makes the subject unsuitable for the study.
* Have a history of malignant neoplasm within the last 5 years, except for adequately treated cancers of the skin (basal or squamous cell) or carcinoma in situ of the uterine cervix.
* Have required management of acute or chronic infections, as follows:

  * Currently on any suppressive therapy for a chronic infection (such as tuberculosis, pneumocystis, cytomegalovirus, herpes simplex virus, herpes zoster, and atypical mycobacteria).
  * Hospitalization for treatment of infection within 60 days of Day 0.
  * Use of parenteral (IV or intramuscular [IM]) antibiotics (antibacterials, antivirals, anti-fungals, or anti-parasitic agents) within 60 days of Day 0.
* Subjects who have evidence of serious suicide risk including any history of suicidal behavior in the last 6 months and/or any suicidal ideation of type 4 or 5 on the screening Columbia-Suicide Severity Rating Scale (C-SSRS) in the last 2 months or who, in the investigator's opinion, pose a significant suicide risk.
* Have current drug or alcohol abuse or dependence, or a history of drug or alcohol abuse or dependence within 364 days prior to Day 0.
* Have a historically positive test or test positive at screening for human immunodeficiency virus (HIV) antibody, hepatitis B surface antigen (HBsAg), hepatitis B core antibody, or hepatitis C antibody.
* Have an immunoglobulin (Ig)A deficiency (IgA level < 10 mg/dL).
* Have a grade 3 or greater laboratory abnormality based on the adverse event
* Severity grading tables except for the following that are allowed:

  * Stable grade 3 prothrombin time (PT) secondary to anticoagulant, e.g., warfarin, treatment.
  * Stable grade 3 partial thromboplastin time (PTT) due to lupus anticoagulant and not related to liver disease or anti-coagulant therapy.
  * Stable grade 3/4 proteinuria (<=6 grams/24 hour equivalent by spot urine protein to creatinine ratio allowed).
  * Stable grade 3 hypoalbuminemia due to lupus nephritis, and not related to liver disease or malnutrition.
  * Stable grade 3 gamma glutamyl transferase (GGT) elevation due to lupus hepatitis, and not related to alcoholic liver disease, uncontrolled diabetes, or viral hepatitis. If present, any abnormalities in alanine transaminase (ALT) and/or aspartate transaminase (AST) must be <=grade 2.
  * Stable grade 3 hemoglobin reduction due to lupus.
  * Stable grade 3 neutropenia or stable grade 3 white blood cell count.
* Have a history of an anaphylactic reaction to parenteral administration of contrast agents, human or murine proteins, or monoclonal antibodies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 503 (Actual)
Dates: Start 2013-02-19 (Actual); Primary Completion 2018-06-18 (Actual); Study Completion 2019-01-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (76):
- United States (52):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Covina, California
  - GSK Investigational Site, La Palma, California
  - GSK Investigational Site, Lakewood, California
  - GSK Investigational Site, Los Alamitos, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Murrieta, California
  - GSK Investigational Site, Upland, California
  - GSK Investigational Site, Bridgeport, Connecticut
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Aventura, Florida
  - GSK Investigational Site, DeBary, Florida
  - GSK Investigational Site, Fort Lauderdale, Florida
  - GSK Investigational Site, Longwood, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Miami Lakes, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Plantation, Florida
  - GSK Investigational Site, Tamarac, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Duluth, Georgia
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Baton Rouge, Louisiana
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Detroit, Michigan
  - GSK Investigational Site, Lansing, Michigan
  - GSK Investigational Site, Jackson, Mississippi
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Clifton, New Jersey
  - GSK Investigational Site, Brooklyn, New York
  - GSK Investigational Site, Great Neck, New York
  - GSK Investigational Site, Manhasset, New York
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Chapel Hill, North Carolina
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Greenville, North Carolina
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Wilmington, North Carolina
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Wyomissing, Pennsylvania
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Columbia, South Carolina
  - GSK Investigational Site, Jackson, Tennessee
  - GSK Investigational Site, Memphis, Tennessee
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, The Woodlands, Texas
  - GSK Investigational Site, Arlington, Virginia
- Brazil (11):
  - GSK Investigational Site, Salvador, Estado de Bahia
  - GSK Investigational Site, Cuiabá, Mato Grosso
  - GSK Investigational Site, Juiz de Fora, Minas Gerais
  - GSK Investigational Site, Curitba, Paraná
  - GSK Investigational Site, Porto Alegre, Rio Grande do Sul
  - GSK Investigational Site, Campinas, São Paulo
  - GSK Investigational Site, Santo André, São Paulo
  - GSK Investigational Site, Belo Horizonte, Minas Gerais
  - GSK Investigational Site, Campo Grande
  - GSK Investigational Site, Rio de Janeiro
  - GSK Investigational Site, São Paulo
- Colombia (4):
  - GSK Investigational Site, Barranquilla
  - GSK Investigational Site, Bucaramanga
  - GSK Investigational Site, Cali
  - GSK Investigational Site, Medellín
- France (2):
  - GSK Investigational Site, Fort de France
  - GSK Investigational Site, Paris
- South Africa (4):
  - GSK Investigational Site, Durban, KwaZulu-Natal
  - GSK Investigational Site, Diepkloof
  - GSK Investigational Site, Johannesburg
  - GSK Investigational Site, Panorama / Cape Town
- United Kingdom (3):
  - GSK Investigational Site, Basildon, Essex
  - GSK Investigational Site, London
  - GSK Investigational Site, Manchester

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study is available via the Clinical Study Data Request site
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (copy the URL below to your browser)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://www.clinicalstudydatarequest.com/Posting.aspx?ID=20862

REFERENCES:
- [Background] Ginzler E, Guedes Barbosa LS, D'Cruz D, Furie R, Maksimowicz-McKinnon K, Oates J, Santiago MB, Saxena A, Sheikh S, Bass DL, Burriss SW, Gilbride JA, Groark JG, Miller M, Pierce A, Roth DA, Ji B. Phase III/IV, Randomized, Fifty-Two-Week Study of the Efficacy and Safety of Belimumab in Patients of Black African Ancestry With Systemic Lupus Erythematosus. Arthritis Rheumatol. 2022 Jan;74(1):112-123. doi: 10.1002/art.41900. Epub 2021 Dec 9. PMID 34164944
- [Derived] Nikolopoulos D, Cetrez N, Lindblom J, Parodis I. Neuropsychiatric involvement in systemic lupus erythematosus contributes to organ damage beyond the nervous system: a post-hoc analysis of 5 phase III randomized clinical trials. Rheumatol Int. 2024 Sep;44(9):1679-1689. doi: 10.1007/s00296-024-05667-5. Epub 2024 Aug 8. PMID 39115551
- [Derived] Arends EJ, Zlei M, Tipton CM, Cotic J, Osmani Z, de Bie FJ, Kamerling SWA, van Maurik A, Dimelow R, Gregan YI, Fox NL, Rabelink TJ, Roth DA, Sanz I, van Dongen JJM, van Kooten C, Teng YKO. Disruption of memory B-cell trafficking by belimumab in patients with systemic lupus erythematosus. Rheumatology (Oxford). 2024 Sep 1;63(9):2387-2398. doi: 10.1093/rheumatology/keae286. PMID 38775637
- [Derived] Brunner HI, Abud-Mendoza C, Mori M, Pilkington CA, Syed R, Takei S, Viola DO, Furie RA, Navarra S, Zhang F, Bass DL, Eriksson G, Hammer AE, Ji BN, Okily M, Roth DA, Quasny H, Ruperto N. Efficacy and safety of belimumab in paediatric and adult patients with systemic lupus erythematosus: an across-study comparison. RMD Open. 2021 Sep;7(3):e001747. doi: 10.1136/rmdopen-2021-001747. PMID 34531304

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study evaluated the efficacy and safety of belimumab compared with placebo in adult participants with Systemic Lupus Erythematosus (SLE). This was a multicenter study conducted at United States (88 centers), United Kingdom (6), South Africa (5), France (4), Columbia (6) and Brazil (18).
Pre-assignment Details: A total of 503 participants were randomized of which 496 received at-least one dose of study medication during double-blinded phase (7 participants were randomized but not treated as they were randomized in error). A total of 359 out of 373 participants who completed double-blinded phase opted to continue optional open-label (OL) extension phase.
Groups:
- Placebo to Belimumab 10 mg/kg: In double-blinded phase, participants received matching placebo to belimumab administered as intravenous (IV) infusion plus standard of care through 52 weeks. In open-label phase, participants received belimumab 10 milligram per kilogram (mg/kg) administered as IV infusion plus standard of care every 28 days from Week 52 through Week 76.
- Belimumab 10 mg/kg to Belimumab 10 mg/kg: In double-blinded phase, participants received belimumab 10 mg/kg administered as IV infusion plus standard of care through 52 weeks. In open-label phase, participants received belimumab 10 mg/kg administered as IV infusion plus standard of care every 28 days from Week 52 through Week 76.
Period: Double-blinded (Up to Week 52)
Arm/Group | Placebo to Belimumab 10 mg/kg | Belimumab 10 mg/kg to Belimumab 10 mg/kg
Started | 165 | 331
Completed | 121 | 252
Not Completed | 44 | 79
Not completed — Site Closed | 3 | 5
Not completed — Protocol Violation | 2 | 6
Not completed — Lost to Follow-up | 1 | 8
Not completed — Physician Decision | 9 | 12
Not completed — Lack of Efficacy | 9 | 15
Not completed — Withdrawal by Subject | 10 | 14
Not completed — Adverse Event | 10 | 19
Period: Open-label (Week 52 to Week 76)
Arm/Group | Placebo to Belimumab 10 mg/kg | Belimumab 10 mg/kg to Belimumab 10 mg/kg
Started | 117 (As the OL phase was optional, participants did not choose to enter the OL Phase.) | 242 (As the OL phase was optional, participants did not choose to enter the OL Phase.)
Completed | 107 | 220
Not Completed | 10 | 22
Not completed — Withdrawal by Subject | 5 | 2
Not completed — Physician Decision | 1 | 4
Not completed — Lost to Follow-up | 1 | 4
Not completed — Site Closed | 2 | 8
Not completed — Protocol Violation | 0 | 2
Not completed — Lack of Efficacy | 0 | 2
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo to Belimumab 10 mg/kg | Belimumab 10 mg/kg to Belimumab 10 mg/kg | Total
Number analyzed (Participants) | 165 | 331 | 496
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39.5 (12.06) | 38.7 (11.00) | 38.9 (11.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 158 | 322 | 480
  Male | 7 | 9 | 16
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Black or African American | 165 | 331 | 496

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving a Systemic Lupus Erythematosus Responder Index (SRI) Response Rate With the Modified Systemic Lupus Erythematosus Disease Activity Index- 2K (SLEDAI-2K) Scoring for Proteinuria at Week 52 [DB Phase]
Description: SRI response is defined as >=4 point reduction, from Baseline in safety of estrogen in Lupus National Assessment(SELENA)SLEDAI[SS] score (with modified SLEDAI-2K scoring for proteinuria [PU]), no worsening (increase of <0.30 points from Baseline) in Physician's Global Assessment (PGA) and no new British Isles Lupus Assessment Group of SLE clinics(BILAG)A organ domain score [ODS] or 2 new BILAG B ODS compared with Baseline. Drop-outs and treatment failures were set to non-responders. Analysis performed using a logistic regression model for comparison between belimumab and placebo with covariates treatment group, Baseline SS score (with modified SLEDAI-2K scoring for PU) (<=9 versus [vs.] >=10), Baseline complement levels (low C3 and/or C4 vs. no low C3 or C4) and region (United States [US]/Canada vs. Rest of World). The Modified Intention-To-Treat (mITT) population comprised of safety population excluding participants who had any assessment at 3 sites (202196, 202513 or 107286).
Time Frame: Week 52
Population: mITT Population. One participant in the mITT population Belimumab 10 mg/kg arm did not have a screening or Baseline PGA assessment; therefore, this participant did not contribute to the SRI/component analysis.
Measure: Number; unit: Percentage of participants
Groups:
- Placebo (DB Phase): In DB phase, participants received matching placebo to belimumab administered as IV infusion plus standard of care through 52 weeks.
- Belimumab 10 mg/kg (DB Phase): In DB phase, participants received belimumab 10 mg/kg administered as IV infusion plus standard of care through 52 weeks.
Arm/Group | Placebo (DB Phase) | Belimumab 10 mg/kg (DB Phase)
Number analyzed (Participants) | 149 | 298
Percentage of participants | 41.6 | 48.7
Statistical Analysis 1: Comparison: Placebo (DB Phase) vs Belimumab 10 mg/kg (DB Phase); Test type: Superiority; p = 0.1068, Regression, Logistic; Odds Ratio (OR) = 1.40, 95% CI 2-sided [0.93 to 2.11]

2. Primary Outcome: Percentage of Participants Achieving a SRI Response Rate With the Modified SLEDAI-2K Scoring for Proteinuria at Week 24 of OL Phase
Description: SRI response is defined as >=4 point reduction, from OL Baseline in SS score (with the modified SLEDAI-2K scoring for PU), no worsening (increase of <0.30 points from OL Baseline) in PGA and no new BILAG A ODS or 2 new BILAG B ODS compared with OL Baseline. For participants switching from placebo to belimumab 10 mg/kg IV in the OL phase, Baseline was defined as the last assessment at the end of the double-blind phase (i.e. Week 52) pre-OL treatment. For participants that received belimumab 10 mg/kg IV during the double-blind phase and continued to receive belimumab 10 mg/kg IV during the OL phase, Baseline was defined as Day 1 of the double-blind phase.
Time Frame: Week 24 of OL phase (Week 76)
Population: mITT OL population comprised of Intent-to-Treat (ITT) OL population (all randomized participants who received at least one dose of OL treatment) excluding participants who had any assessment at 3 sites (202196, 202513 or 107286). Only those participants with data available at the specified data points were analyzed.
Measure: Number; unit: Percentage of participants
Groups:
- Placebo to Belimumab 10 mg/kg (OL Phase); Belimumab 10 mg/kg to Belimumab 10 mg/kg (OL Phase): In OL phase, participants received belimumab 10 mg/kg administered as IV infusion plus standard of care every 28 days from Week 52 through Week 76
Arm/Group | Placebo to Belimumab 10 mg/kg (OL Phase) | Belimumab 10 mg/kg to Belimumab 10 mg/kg (OL Phase)
Number analyzed (Participants) | 69 | 208
Percentage of participants | 18.8 | 73.6

3. Primary Outcome: Number of Participants With Non-serious Adverse Events (nSAEs) and Serious Adverse Event (SAEs) [OL Phase]
Description: An adverse event (AE) is any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAE is defined as any untoward medical occurrence that; results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, other situations judged by physician, is associated with liver injury and impaired liver function. Number of participants who had common nSAEs (>=5%) and any SAEs are presented. For Safety, participants that completed DB and OL phase, an additional 8 weeks follow-up was conducted (Week 84).
Time Frame: Week 52 to Week 84
Population: Intent-to-Treat (ITT) OL Population comprised of all randomized participants who received atleast one dose of open label treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo to Belimumab 10 mg/kg (OL Phase) | Belimumab 10 mg/kg to Belimumab 10 mg/kg (OL Phase)
Number analyzed (Participants) | 117 | 242
Participants
  nSAEs | 23 | 49
  SAEs | 6 | 13

4. Primary Outcome: Number of Participants With Severe AEs [OL Phase]
Description: An AE is any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Number of participants with severe AEs have been presented. For Safety, participants that completed DB and OL phase, an additional 8 weeks follow-up was conducted (Week 84).
Time Frame: Week 52 to Week 84
Population: ITT OL Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo to Belimumab 10 mg/kg (OL Phase) | Belimumab 10 mg/kg to Belimumab 10 mg/kg (OL Phase)
Number analyzed (Participants) | 117 | 242
Participants | 10 | 9

5. Primary Outcome: Number of Participants With AEs Leading to Treatment Discontinuation [OL Phase]
Description: An AE is any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Number of participants with AEs leading to treatment discontinuation have been presented. For Safety, participants that completed DB and OL phase, an additional 8 weeks follow-up was conducted (Week 84).
Time Frame: Week 52 to Week 84
Population: ITT OL Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo to Belimumab 10 mg/kg (OL Phase) | Belimumab 10 mg/kg to Belimumab 10 mg/kg (OL Phase)
Number analyzed (Participants) | 117 | 242
Participants | 1 | 0

6. Primary Outcome: Number of Participants With Worst Toxicity Grade 3 or 4 for Hematology Parameters [OL Phase]
Description: Blood samples were collected for the assessment of hematology parameters. The parameters assessed were activated partial thromboplastin time (APTT), hemoglobin, leukocytes, neutrophils, platelets and prothrombin time. Grading was assigned as mild (Grade 1), moderate (grade 2), severe (Grade 3) and potentially life-threatening (Grade 4) according to Division of Microbiology and Infectious Diseases (DMID [Modified from DMID Adult Toxicity Tables, 2001]) AE Severity Grading. Number of participants with worst toxicity Grade 3 or 4 for hematology parameters have been presented. For Safety, participants that completed DB and OL phase, an additional 8 weeks follow-up was conducted (Week 84).
Time Frame: Week 52 to Week 84
Population: ITT OL Population. Only those participants with data available at the specified data points were analyzed (represented by n=X in the category titles).
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo to Belimumab 10 mg/kg (OL Phase) | Belimumab 10 mg/kg to Belimumab 10 mg/kg (OL Phase)
Number analyzed (Participants) | 115 | 235
Participants
  APTT, Grade 3, n=93,203: number analyzed (Participants) | 93 | 203
  APTT, Grade 3, n=93,203 | 0 | 1
  APTT, Grade 4, n=93,203: number analyzed (Participants) | 93 | 203
  APTT, Grade 4, n=93,203 | 0 | 0
  Hemoglobin, Grade 3, n=115,235 | 4 | 6
  Hemoglobin, Grade 4, n=115,235 | 0 | 0
  Leukocytes, Grade 3, n=114,235: number analyzed (Participants) | 114 | 235
  Leukocytes, Grade 3, n=114,235 | 0 | 6
  Leukocytes, Grade 4, n=114,235: number analyzed (Participants) | 114 | 235
  Leukocytes, Grade 4, n=114,235 | 0 | 0
  Neutrophils, Grade 3, n=114,234: number analyzed (Participants) | 114 | 234
  Neutrophils, Grade 3, n=114,234 | 2 | 6
  Neutrophils, Grade 4, n=114,234: number analyzed (Participants) | 114 | 234
  Neutrophils, Grade 4, n=114,234 | 0 | 1
  Platelets, Grade 3, n=115,235 | 0 | 0
  Platelets, Grade 4, n=115,235 | 0 | 0
  Prothrombin time, Grade 3, n=93, 204: number analyzed (Participants) | 93 | 204
  Prothrombin time, Grade 3, n=93, 204 | 3 | 2
  Prothrombin time, Grade 4, n=93, 204: number analyzed (Participants) | 93 | 204
  Prothrombin time, Grade 4, n=93, 204 | 1 | 3

7. Primary Outcome: Number of Participants With Worst Toxicity Grade of 3 or 4 for Clinical Chemistry Parameters [OL Phase]
Description: Blood samples were collected for the assessment of liver function and other chemistry parameters. The parameters assessed were alkaline phosphatase (ALP), alanine aminotransferase (ALT), aspartate aminotransferase (AST), gamma glutamyl transferase (GGT), bilirubin, albumin, creatinine, hyperglycemia, hypoglycemia and urate. Grading was assigned as mild (Grade 1), moderate (grade 2), severe (Grade 3) and potentially life-threatening (Grade 4) according to DMID AE Severity Grading. Number of participants with worst toxicity Grade of 3 or 4 for liver function and other chemistry parameters have been presented. For Safety, participants that completed DB and OL phase, an additional 8 weeks follow-up was conducted (Week 84).
Time Frame: Week 52 to Week 84
Population: ITT OL Population. Only those participants with data available at the specified data points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo to Belimumab 10 mg/kg (OL Phase) | Belimumab 10 mg/kg to Belimumab 10 mg/kg (OL Phase)
Number analyzed (Participants) | 115 | 236
Participants
  ALP, Grade 3 | 0 | 0
  ALP, Grade 4 | 0 | 0
  ALT, Grade 3 | 0 | 0
  ALT, Grade 4 | 0 | 0
  AST, Grade 3 | 0 | 0
  AST, Grade 4 | 0 | 0
  Bilirubin, Grade 3 | 0 | 0
  Bilirubin, Grade 4 | 0 | 0
  GGT, Grade 3 | 0 | 1
  GGT, Grade 4 | 0 | 0
  Albumin, Grade 3 | 0 | 2
  Albumin, Grade 4 | 1 | 0
  Creatinine, Grade 3 | 0 | 0
  Creatinine, Grade 4 | 0 | 0
  Hypoglycemia, Grade 3 | 0 | 0
  Hypoglycemia, Grade 4 | 0 | 0
  Hyperglycemia, Grade 3 | 1 | 4
  Hyperglycemia, Grade 4 | 0 | 0
  Urate, Grade 3 | 0 | 0
  Urate, Grade 4 | 0 | 0

8. Primary Outcome: Number of Participants With Worst Toxicity Grade of 3 or 4 for Urinalysis Parameters [OL Phase]
Description: Urinalysis parameters assessed were urine protein and protein/creatinine. Urine samples were collected for the measurement of urinalysis parameters by dipstick method. Grading was assigned as mild (Grade 1), moderate (grade 2), severe (Grade 3) and potentially life-threatening (Grade 4) according to DMID AE Severity Grading. Number of participants with worst toxicity grade of 3 or 4 for urinalysis parameters have been presented. For Safety, participants that completed DB and OL phase, an additional 8 weeks follow-up was conducted (Week 84).
Time Frame: Week 52 to Week 84
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo to Belimumab 10 mg/kg (OL Phase) | Belimumab 10 mg/kg to Belimumab 10 mg/kg (OL Phase)
Number analyzed (Participants) | 115 | 234
Participants
  Protein, Grade 3, n=115, 234 | 0 | 0
  Protein, Grade 4, n=115,234 | 0 | 0
  Protein/Creatinine, Grade 3,n=112,227: number analyzed (Participants) | 112 | 227
  Protein/Creatinine, Grade 3,n=112,227 | 5 | 5
  Protein/Creatinine, Grade 4, n=112,227: number analyzed (Participants) | 112 | 227
  Protein/Creatinine, Grade 4, n=112,227 | 3 | 0

9. Primary Outcome: Number of Participants With Worst Toxicity Grade of 3 or 4 of Immunoglobulins [OL Phase]
Description: Serum samples were obtained for the measurement of immunoglobulin G. Grading was assigned as mild (Grade 1), moderate (grade 2), severe (Grade 3) and potentially life threatening (Grade 4) according to DMID AE Severity Grading. Number of participants with worst toxicity grade of 3 or 4 of immunoglobulin G have been presented. For Safety, participants that completed DB and OL phase, an additional 8 weeks follow-up was conducted (Week 84).
Time Frame: Week 52 to Week 84
Population: ITT OL Population. Only those participants with data available at the specified data points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo to Belimumab 10 mg/kg (OL Phase) | Belimumab 10 mg/kg to Belimumab 10 mg/kg (OL Phase)
Number analyzed (Participants) | 117 | 239
Participants
  Grade 3 | 0 | 1
  Grade 4 | 0 | 0

10. Secondary Outcome: Percentage of Participants Achieving SRI-SS Response Rate at Week 52 [DB Phase]
Description: SRI is defined as >=4 point reduction, from Baseline in SS score, no worsening (increase of <0.30 points from Baseline) in PGA and no new BILAG A organ domain score or 2 new BILAG B organ domain scores compared with Baseline. Drop-outs and Treatment failures were set to non-responders. Analysis was performed using a logistic regression model for the comparison between belimumab and placebo with covariates treatment group, Baseline SS score (<=9 vs. >=10), Baseline complement levels (low C3 and/or C4 vs. no low C3 or C4) and region (US/Canada vs. Rest of World).
Time Frame: Week 52
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo (DB Phase) | Belimumab 10 mg/kg (DB Phase)
Number analyzed (Participants) | 149 | 298
Percentage of participants | 41.6 | 49.0
Statistical Analysis 1: Comparison: Placebo (DB Phase) vs Belimumab 10 mg/kg (DB Phase); Test type: Superiority; p = 0.0937, Regression, Logistic — Nominal p-value due to step-down sequential testing procedure; Odds Ratio (OR) = 1.42, 95% CI 2-sided [0.94 to 2.15]

11. Secondary Outcome: Percentage of Participants Achieving SRI-SS Response Rate With the SELENA SLEDAI for Scoring of Proteinuria at Week 24 of OL Phase
Description: SRI response is defined as >=4 point reduction, from OL Baseline in SS scoring for PU, no worsening (increase of <0.30 points from OL Baseline) in PGA and no new BILAG A ODS or 2 new BILAG B ODS compared with OL Baseline. For participants switching from placebo to belimumab 10 mg/kg IV in the open-label phase, Baseline was defined as the last assessment at the end of the double-blind phase (i.e. Week 52) pre-OL treatment. For participants that received belimumab 10 mg/kg IV during the double-blind phase and continued to receive belimumab 10 mg/kg IV during the open-label phase, Baseline was defined as Day 1 of the double-blind phase.
Time Frame: Week 24 of OL phase (Week 76)
Population: mITT OL Population. Only those participants with data available at the specified data points were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo to Belimumab 10 mg/kg (OL Phase) | Belimumab 10 mg/kg to Belimumab 10 mg/kg (OL Phase)
Number analyzed (Participants) | 67 | 208
Percentage of participants | 19.4 | 73.1

12. Secondary Outcome: Time to First Severe Flare (as Measured by the Modified SLE Flare Index) up to 52 Weeks [DB Phase]
Description: Time to first severe SLE flare is defined as the number of days from treatment start date until the participant met an event (event date - treatment start date +1). Analyses of severe SLE flare was performed on modified SS SLE flare index that excludes severe flares (SF) that were triggered only by an increase in SS score to >12 (this may only represent a modest increase in disease activity). Treatment failures were imputed as SF. For participants who died, data were censored at date of death if no SF occurred before death. Only post-Baseline SF were considered. Analysis was performed using Cox proportional hazards model for the comparison between belimumab and placebo adjusting for Baseline SS-S2K score (<=9 vs. >=10), baseline complement levels (at least 1 C3/C4 low vs. no C3/C4 low), and region (US/Canada vs. Rest of World). Median and inter-Quartile range (1st and 3rd Quartiles) have been presented.
Time Frame: Up to 52 Weeks
Population: mITT Population
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Placebo (DB Phase) | Belimumab 10 mg/kg (DB Phase)
Number analyzed (Participants) | 149 | 299
Days | NA [346 to NA] — NA indicated data was not available because the number of events was too low to estimate the value. | NA [NA to NA] — NA indicated data was not available because the number of events was too low to estimate the value.
Statistical Analysis 1: Comparison: Placebo (DB Phase) vs Belimumab 10 mg/kg (DB Phase); Test type: Superiority; p = 0.2264, Cox proportional hazards model — Nominal p-value due to step-down sequential testing procedure; Hazard Ratio (HR) = 0.77, 95% CI 2-sided [0.51 to 1.17]

13. Secondary Outcome: Time to First Severe Flare (as Measured by the Modified SLE Flare Index) [OL Phase]
Description: Time to first severe SLE flare is defined as the number of days from OL treatment start date until the participant met an event (event date - OL treatment start date +1). Analyses of severe SLE flare was performed on modified SS SLE flare index that excludes SF that were triggered only by an increase in SS score to >12. For participants who died, data were censored at date of death if no SF occurred before death. Only post first OL treatment SF were considered. Median and inter-Quartile range (25th and 75th percentile) have been presented.
Time Frame: Up to Week 24 of OL Phase (Week 76)
Population: mITT OL Population
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Placebo to Belimumab 10 mg/kg (OL Phase) | Belimumab 10 mg/kg to Belimumab 10 mg/kg (OL Phase)
Number analyzed (Participants) | 109 | 225
Days | NA [NA to NA] — NA indicated data was not available because the number of events was too low to estimate the value. | 232 [232 to NA] — NA indicated data was not available because the number of events was too low to estimate the value.

14. Secondary Outcome: Percent of Participants Whose Average Prednisone Dose Had Been Reduced by >=25% From Baseline to <=7.5 mg/Day During Week 40 Through 52, in Participants Receiving Greater Than 7.5 mg/Day at Baseline [DB Phase]
Description: Average (avg.) daily prednisone (PRED.) dose was calculated taking into account all steroids taken intravenously, intramuscularly, subcutaneously, intradermally and orally for both Systemic Lupus Erythema (SLE) and non-SLE reasons. A responder was defined as having a PRED. reduction [REDN.] by >=25% from Baseline to <=7.5 mg/day during Weeks 40 through 52. Drop-outs and Treatment failures were imputed as having no REDN. in PRED. (if Baseline PRED. >7.5 mg/day). At Baseline, the avg. daily prednisone dose [PD] was the sum of all PDs over 7 consecutive days [excluding Day 0], divided (DIV.) by 7. For analysis, the avg. PD was the total PD during Weeks 40 through 52 DIV. by the number of days during Weeks 40 through 52. Analysis was performed using a logistic regression model with covariates treatment group, Baseline PD, Baseline SS-S2K score, (<=9 vs >=10), Baseline complement levels (low C3 and/or C4 vs. no low C3 or C4) and region (US/Canada vs. Rest of World).
Time Frame: Baseline and Week 40 through Week 52
Population: mITT Population. Only participants with Baseline prednisone dose >7.5 mg/day were included.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo (DB Phase) | Belimumab 10 mg/kg (DB Phase)
Number analyzed (Participants) | 95 | 184
Percentage of participants | 12.6 | 14.7
Statistical Analysis 1: Comparison: Placebo (DB Phase) vs Belimumab 10 mg/kg (DB Phase); Test type: Superiority; p = 0.4996, Regression, Logistic — Nominal p-value due to step-down sequential testing procedure; Odds Ratio (OR) = 1.30, 95% CI 2-sided [0.61 to 2.80]

15. Secondary Outcome: Percent of Participants Whose Average Prednisone Dose Had Been Reduced to <=7.5 mg/Day in Participants Receiving Greater Than 7.5 mg/Day at Pre-belimumab Baseline (at Week 28 of OL Phase)
Description: Average daily prednisone dose was calculated taking into account all steroids taken intravenously, intramuscularly, subcutaneously, intradermally and orally for both SLE and non-SLE reasons. A responder was defined as a participant who decreased their daily prednisone dose to <=7.5 mg/day from an OL Baseline dose >7.5 mg/day. The OL Baseline was defined as the last available value prior to the initiation of treatment with belimumab. The average daily prednisone dose was the sum of all PDs over 7 consecutive days including OL Week 28 divided by 7. Only those participants with data available at the specified data points were analyzed.
Time Frame: OL Baseline and Week 28 of OL Phase (Week 80)
Population: mITT OL Population. Only those participants with data available at the specified data points were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo to Belimumab 10 mg/kg (OL Phase) | Belimumab 10 mg/kg to Belimumab 10 mg/kg (OL Phase)
Number analyzed (Participants) | 54 | 138
Percentage of participants | 14.8 | 31.9

16. Secondary Outcome: Number of Participants With nSAEs and SAEs [DB Phase]
Description: An AE is any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. A SAE is defined as any untoward medical occurrence that; results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, other situations judged by physician, is associated with liver injury and impaired liver function. Safety population was defined as all participants who were randomized and treated with at least one dose of study treatment. Number of participants who had common nSAEs (>=5%) and any SAEs are presented.
Time Frame: Up to 52 Weeks
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (DB Phase) | Belimumab 10 mg/kg (DB Phase)
Number analyzed (Participants) | 165 | 331
Participants
  nSAE | 77 | 196
  SAE | 31 | 36

17. Secondary Outcome: Number of Participants With Severe AEs [DB Phase]
Description: An AE is any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Number of participants with severe AEs have been presented.
Time Frame: Up to 52 Weeks
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (DB Phase) | Belimumab 10 mg/kg (DB Phase)
Number analyzed (Participants) | 165 | 331
Participants | 37 | 46

18. Secondary Outcome: Number of Participants With AEs Leading to Treatment Discontinuation [DB Phase]
Description: An AE is any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Number of participants with AEs leading to treatment discontinuation have been presented.
Time Frame: Up to 52 Weeks
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (DB Phase) | Belimumab 10 mg/kg (DB Phase)
Number analyzed (Participants) | 165 | 331
Participants | 12 | 22

19. Secondary Outcome: Number of Participants With Worst Toxicity Grade 3 or 4 for Hematology Parameters [DB Phase]
Description: Blood samples were collected for the assessment of hematology parameters up to 52 Weeks. The parameters assessed were APTT, hemoglobin, leukocytes, neutrophils, platelets and prothrombin time. Grading was assigned as mild (Grade 1), moderate (grade 2), severe (Grade 3) and potentially life threatening according to DMID AE Severity Grading. Number of participants with worst toxicity Grade of 3 or 4 for hematology parameters have been presented.
Time Frame: Up to 52 weeks
Population: Safety Population. Only those participants with data available at the specified data points were analyzed (represented by n=X in the category titles).
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (DB Phase) | Belimumab 10 mg/kg (DB Phase)
Number analyzed (Participants) | 161 | 327
Participants
  APTT, Grade 3, n=159,318: number analyzed (Participants) | 159 | 318
  APTT, Grade 3, n=159,318 | 0 | 3
  APTT, Grade 4, n=159,318: number analyzed (Participants) | 159 | 318
  APTT, Grade 4, n=159,318 | 0 | 2
  Hemoglobin, Grade 3, n=161,327 | 5 | 15
  Hemoglobin, Grade 4, n=161,327 | 1 | 0
  Leukocytes, Grade 3, n=161,327 | 3 | 17
  Leukocytes, Grade 4, n=161,327 | 1 | 0
  Neutrophils, Grade 3, n=161,327 | 9 | 28
  Neutrophils, Grade 4, n=161,327 | 1 | 5
  Platelets, Grade 3, n=161,327 | 1 | 1
  Platelets, Grade 4, n=161,327 | 0 | 1
  Prothrombin time, Grade 3, n=159, 318: number analyzed (Participants) | 159 | 318
  Prothrombin time, Grade 3, n=159, 318 | 8 | 10
  Prothrombin time, Grade 4, n=159,318: number analyzed (Participants) | 159 | 318
  Prothrombin time, Grade 4, n=159,318 | 2 | 6

20. Secondary Outcome: Number of Participants With Worst Toxicity Grade of 3 or 4 for Clinical Chemistry Parameters [DB Phase]
Description: Blood samples were collected for the assessment of liver function and other chemistry parameters up to 52 Weeks. The parameters assessed were ALT, AST, GGT, albumin, hyperglycemia and hypoglycemia. Grading was assigned as mild (Grade 1), moderate (grade 2), severe (Grade 3) and potentially life threatening according to DMID AE Severity Grading. Only those participants with worst toxicity Grade of 3 or 4 for other chemistry parameters have been presented.
Time Frame: Up to 52 weeks
Population: Safety Population. Only those participants with data available at the specified data points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (DB Phase) | Belimumab 10 mg/kg (DB Phase)
Number analyzed (Participants) | 161 | 327
Participants
  ALT, Grade 3 | 0 | 2
  AST, Grade 3 | 0 | 2
  GGT, Grade 3 | 6 | 6
  GGT, Grade 4 | 0 | 1
  Albumin, Grade 3 | 5 | 3
  Albumin, Grade 4 | 1 | 1
  Hyperglycemia, Grade 3 | 4 | 7
  Hyperglycemia, Grade 4 | 1 | 1
  Hypoglycemia, Grade 3 | 0 | 4
  Hypoglycemia, Grade 4 | 3 | 1

21. Secondary Outcome: Number of Participants With Worst Toxicity Grade of 3 or 4 for Urinalysis Parameters [DB Phase]
Description: Urinalysis parameters assessed were urine protein and protein/creatinine. Urine samples were collected for the measurement of urinalysis parameters by dipstick method up to 52 Weeks. Grading was assigned as mild (Grade 1), moderate (grade 2), severe (Grade 3) and potentially life threatening according to DMID AE Severity Grading. Only those participants with worst toxicity grade of 3 or 4 for urinalysis parameters have been presented.
Time Frame: Up to 52 weeks
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (DB Phase) | Belimumab 10 mg/kg (DB Phase)
Number analyzed (Participants) | 161 | 324
Participants
  Protein, Grade 3, n=161, 324 | 0 | 1
  Protein/creatinine, Grade 3,n=161,322: number analyzed (Participants) | 161 | 322
  Protein/creatinine, Grade 3,n=161,322 | 8 | 25
  Protein/creatinine, Grade 4, n=161,322: number analyzed (Participants) | 161 | 322
  Protein/creatinine, Grade 4, n=161,322 | 12 | 11

ADVERSE EVENTS:
Time Frame: nSAEs and SAEs were collected from the start of study treatment up to Week 52 for Double Blind phase and from Week 52 to Week 84 for the Open Label phase. Participants that completed DB and OL phase, an additional 8 weeks follow-up was conducted (Week 84).
Description: nSAEs and SAEs were reported for the Safety Population which comprised of all randomized participants who received at least 1 dose of study treatment for Double Blind phase and ITT OL Population which comprised of all randomized participants who received at least 1 dose of OL treatment for OL phase.
Arm/Group | Placebo (DB Phase) | Belimumab 10 mg/kg (DB Phase) | Placebo to Belimumab 10 mg/kg (OL Phase) | Belimumab 10 mg/kg to Belimumab 10 mg/kg (OL Phase)
All-Cause Mortality (participants affected / at risk) | 0/165 | 2/331 | 0/117 | 0/242
Serious Adverse Events (participants affected / at risk) | 31/165 | 36/331 | 6/117 | 13/242
Other Adverse Events (participants affected / at risk) | 77/165 | 196/331 | 23/117 | 49/242
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (DB Phase) (N=165) | Belimumab 10 mg/kg (DB Phase) (N=331) | Placebo to Belimumab 10 mg/kg (OL Phase) (N=117) | Belimumab 10 mg/kg to Belimumab 10 mg/kg (OL Phase) (N=242)
Pneumonia (Infections and infestations) | 6 (6) | 2 (2) | 0 (0) | 2 (2)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (4) | 0 (0) | 1 (1)
Lupus nephritis (Renal and urinary disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Pericarditis (Cardiac disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
SLE arthritis (Musculoskeletal and connective tissue disorders) | 1 (2) | 2 (2) | 0 (0) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3) | 0 (0) | 1 (1)
Lupus pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Amoebic colitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthritis gonococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Atypical pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Azotaemia (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Butterfly rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coma (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dengue fever (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression suicidal (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dystonia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Glomerulonephritis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Idiopathic intracranial hypertension (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Idiopathic orbital inflammation (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lupus pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lupus vasculitis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malignant hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Meningitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nephrotic syndrome (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Radiculopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Raynaud's phenomenon (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Serositis (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Small intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Soft tissue inflammation (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma of the cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Systemic lupus erythematosus rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vasculitis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Viral tonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Chorea (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hemiparesis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oesophageal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Soft tissue infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (DB Phase) (N=165) | Belimumab 10 mg/kg (DB Phase) (N=331) | Placebo to Belimumab 10 mg/kg (OL Phase) (N=117) | Belimumab 10 mg/kg to Belimumab 10 mg/kg (OL Phase) (N=242)
Upper respiratory tract infection (Infections and infestations) | 14 (20) | 48 (58) | 4 (6) | 20 (21)
Urinary tract infection (Infections and infestations) | 19 (24) | 43 (57) | 7 (7) | 13 (15)
Headache (Nervous system disorders) | 18 (25) | 39 (47) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 17 (23) | 28 (35) | 7 (8) | 16 (18)
Diarrhoea (Gastrointestinal disorders) | 9 (12) | 31 (34) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 9 (9) | 26 (33) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 15 (21) | 18 (29) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 10 (10) | 18 (18) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 10 (12) | 16 (17) | 7 (7) | 3 (3)
Vomiting (Gastrointestinal disorders) | 7 (8) | 19 (21) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 18 (23) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 9 (9) | 15 (15) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 4 (5) | 18 (21) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-02-09): https://cdn.clinicaltrials.gov/large-docs/41/NCT01632241/Prot_000.pdf
  • Statistical Analysis Plan (2019-02-14): https://cdn.clinicaltrials.gov/large-docs/41/NCT01632241/SAP_002.pdf